CLINICAL TRIAL: NCT01072292
Title: Nurse Managed Cognitive Behavioral Therapy for Insomnia in People With Chronic Obstructive Pulmonary Disease
Brief Title: Cognitive Behavioral Therapy for Insomnia in People With Chronic Obstructive Pulmonary Disease(COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Mary C. Kapella, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KO1 NR010749
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT-I (Experimental): CBT-I
  Interventions: Behavioral: CBT-I
- Wellness Education (Active Comparator): Wellness Education
  Interventions: Behavioral: CBT-I

INTERVENTIONS:
Behavioral: CBT-I — CBT-I is a six week program designed to improve sleep quality in people with COPD.

SUMMARY:
A two-phase research study is being conducted. In Phase 1 of the study, the cognitive behavioral therapy intervention for insomnia was implemented in a small (n = 5) group of people with moderate to severe COPD and insomnia. The intervention was pilot-tested to determine feasibility and acceptability, and the intervention will be refined as needed. In Phase 2 of the study, a two-group randomized controlled study (n = 20) will be conducted to test the effects of the cognitive behavioral therapy for insomnia intervention on the primary outcomes of sleep quality and fatigue and the secondary outcomes of mood and functional performance. It is hypothesized that people with COPD receiving cognitive behavioral therapy for insomnia will demonstrate significant improvements in sleep quality, fatigue, mood and functional performance as compared to people with COPD who receive a wellness program. This research will yield valuable information regarding effective interventions aimed at mitigating problems such as poor sleep quality, fatigue and reduced ability to perform valued daily activities. This information will be used to increase the likelihood of long-term successful outcomes such as the ability to maintain productive roles in society for people with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have moderate to severe COPD. Severity of COPD will be defined according to the new GOLD standards (moderate IIA (moderate), 50% < FEV1 < 80% predicted; moderate IIB (severe) 30% < FEV1 < 50%). 58
* Insomnia. Insomnia will be defined as difficulty initiating or maintaining sleep, waking up too early or poor quality sleep. 59
* Subjects must be > 45 years of age with no other major health problems
* Subjects must be clinically stable at the time of enrollment into the study without major exacerbation of COPD within the previous two months.

Exclusion Criteria:

* Evidence of restrictive lung disease or asthma.
* Evidence of a major sleep disorder other than insomnia (sleep apnea evidenced by apnea/hypopnea index of > 10, periodic limb movement disorder, narcolepsy).
* Hypnotic, sedative, anxiolytic or antidepressant use.
* Pulse oximetry (SaO2) reading of < 90% at rest.
* Pulse oximetry (SaO2) reading of < 85% at night for > 5 minutes.
* Significant sleep apnea (apnea/hypopnea index ≥ 10).
* .Acute respiratory infection within the previous 2 months.
* Class > 2 functional status according to the New York Heart Association.
* The presence of a potentially debilitating disease such as cancer, congestive heart failure, kidney disease, liver failure or cirrhosis; evidence of alcohol or drug abuse, musculoskeletal or degenerative nerve disease.
* A self-reported current diagnosis of major depression or psychiatric disease or a Hospital Anxiety and Depression Scale (HADS) depression score of > 11.
* Currently participating in pulmonary rehabilitation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
sleep quality | 6-8 weeks

SECONDARY OUTCOMES:
fatigue/tiredness, using the Chronic Respiratory Disease Questionnaire | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Kapella, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Kapella MC, Herdegen JJ, Perlis ML, Shaver JL, Larson JL, Law JA, Carley DW. Cognitive behavioral therapy for insomnia comorbid with COPD is feasible with preliminary evidence of positive sleep and fatigue effects. Int J Chron Obstruct Pulmon Dis. 2011;6:625-35. doi: 10.2147/COPD.S24858. Epub 2011 Nov 24. PMID 22162648